CLINICAL TRIAL: NCT03514654
Title: Can Patients With Multiple Breast Cancers in the Same Breast Avoid Mastectomy by Having Multiple Lumpectomies to Achieve Equivalent Rates of Local Breast Cancer Recurrence? A Randomised Controlled Feasibility Study.
Brief Title: MIAMI Safe Surgery for Multiple Breast Cancers
Acronym: MIAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/0048
Record Dates: First submitted 2018-03-21; First posted 2018-05-02 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer, Unilateral
Keywords: Breast Cancer; Mastectomy; Therapeutic Mammoplasty; Multiple Ipsilateral Breast Cancers
MeSH Terms: conditions — Unilateral Breast Neoplasms; Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Intervention Model Description: To evaluate whether a sufficient number of eligible patients can be identified and are willing to accept randomisation of the interventions in question. Recruitment and compliance rates of which will inform the feasibility and design of a larger trial
Masking Description: Neither the patients nor the clinical team will be blinded to the trial arms of this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastectomy +/- reconstruction (Active Comparator): Either a simple mastectomy or skin sparing mastectomy technique will be used. Women in this arm will be offered either immediate or delayed breast reconstruction according to standard practice. Reconstructions will be followed by chemotherapy and/or endocrine therapy as determined by local clinicians . Chest wall and/or regional nodal radiotherapy will be prescribed according to local centre policy.
  Interventions: Procedure: Mastectomy
- Therapeutic Mammoplasty (Active Comparator): Therapeutic Mammoplasty (TM) comprises well-established surgical techniques involving volume displacement using breast reduction techniques, or volume replacement to maximize the volume of tissue that can be excised resulting in effective local control whilst maximizing cosmetic outcomes. This group will either have one "disease site" lumpectomy in the case of multifocal tumours or distant "disease site" lumpectomies in multicentric cancers.
  Interventions: Procedure: Therapeutic Mammoplasty

INTERVENTIONS:
Procedure: Mastectomy — Removal of the whole breast.
  Arms: Mastectomy +/- reconstruction
Procedure: Therapeutic Mammoplasty — Excision via lumpectomy of multifocal or multicentric cancers with breast volume displacement techniques to maximise cosmetic outcomes.
  Arms: Therapeutic Mammoplasty

SUMMARY:
Sometimes women have more than one breast cancer in the same breast at the same time. These women are usually offered a mastectomy (removal of that breast) and breast reconstruction. It may be possible to treat these patients by removing each cancer using breast-saving surgery (lumpectomies), used for women with only one breast cancer. Databases show that women who had lumpectomies did well, but they may have been healthier before the surgery than those who had a mastectomy. The investigators need to be sure that lumpectomy is effective, safe, and acceptable for this patient group before making it universally available.

DETAILED DESCRIPTION:
The investigators will run a small study to evaluate whether a sufficient number of eligible patients can be identified and are willing to accept randomisation of the interventions in question. Recruitment and compliance rates of which will inform the feasibility and design of a larger trial. This will comprise a multi-centre randomised controlled trial in women with Multiple Ipsilateral Breast cancer (MIBC) requiring surgery. Participants will receive either Therapeutic Mammoplasty (TM) following excision of each cancer focus or mastectomy (+/- reconstruction). Patients will be randomised (1:1) into either intervention or control group.Therapeutic mammoplasty is an operation to remove breast cancer(s) whilst also significantly reducing the size of the breast. Therapeutic mammoplasty can be used to remove more than one cancer in the breast using separate lumpectomies. Both skin and breast tissue are removed, leaving scars similar to those seen after a standard breast reduction. Each patient is followed up for 12 months post treatment with a total of 50 patients recruited. Timings of the follow-up visits are aligned with standard of care practice for this patient population with quality of life questionnaires and clinical photographs completed before and after surgery. Twenty women will also be invited to an optional semi-structured interview at twelve months.

ELIGIBILITY:
Inclusion Criteria:

1. >40 years with MIBC, with the largest clinical cancer measuring 50mm as part of multifocal or multicentric "disease sites". 50mm may include the size of a single cancer and its surrounding small satellite cancers (6, 7). Clinically diagnosed (ultrasound and biopsy) either axillary lymph node negative or positive where axillary treatment depends on local policy
2. Two disease foci with a minimum of one invasive focus of breast cancer as defined within a "disease site"
3. Suitable for TM (best practice) using one large lumpectomy (multifocal) or any number of "distant" lumpectomies (multicentric) to excise "disease sites"
4. Fit for adjuvant therapy as per pre-operative evaluations (ECG, Chest X-ray, blood biochemistry)
5. Willing and able to provide written informed consent

Exclusion Criteria:

1. Neo-adjuvant therapy
2. Women considered high risk by local centre or known to have BRCA1/2 gene mutation
3. Ductal Carcinoma in situ (DCIS) only, and extensive DCIS
4. Bilateral breast cancers
5. Previous breast cancer (invasive or DCIS in either breast)
6. Pregnancy as confirmed on blood tests or ultrasound examination
7. Metastatic disease
8. Any previous type of breast radiotherapy
9. Significant other clinical risk factors and co-morbidities at the discretion of the treating clinicians
10. Previous or concomitant malignancy except adequately treated: non-melanomatous skin cancer; in situ carcinoma of the cervix and in situ melanoma

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study focuses on female breast cancer
Enrollment: 4 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Number of women screened | 36 Months
  Numbers of women with more than one cancer in the same breast (MIBC) screened for the trial
Number of women eligible for the trial | 36 Months
  Numbers of eligible women based on trial criteria and suitable for therapeutic mammoplasty
Consent rate | 36 Months
  The proportion of women eligible for the trial who provide written informed consent
Compliance with trial procedures | 36 Months
  Rate of compliance with allocated treatment and reason for deviation

SECONDARY OUTCOMES:
Reasons why patients accept or decline randomisation | 36 Months
  Tabulation of reasons why patients accept or decline randomisation (assessed from patient-completed Qualitative Study questionnaire)
Qualitative research (clinical staff) | 36 Months
  Tabulation of views of clinical staff following qualitative interviews
Qualitative research (patients) | 36 Months
  Tabulation of views of participating patients following qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Winters, Principal Investigator — University College, London
Locations (7):
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge
  - South Glasgow Hospitals - New Victoria Hospital / Gartnavel General Hospital, Glasgow
  - Ipswich Hospital, Ipswich
  - St. George's Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Royal Cornwall Hospital, Truro
  - Royal Hampshire Hospital, Winchester

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held on secure servers and will not be released to any third parties until all the main outputs from the studies have been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis by SITU and the Chief Investigator. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Chief Investigator and study group, the sponsor, and funders.

REFERENCES:
- [Derived] Ingram J, Beasant L, Benson J, Brunt AM, Maxwell A, Harvey JR, Greenwood R, Roberts N, Williams N, Johnson D, Winters Z. The challenge of equipoise: qualitative interviews exploring the views of health professionals and women with multiple ipsilateral breast cancer on recruitment to a surgical randomised controlled feasibility trial. Pilot Feasibility Stud. 2022 Feb 28;8(1):46. doi: 10.1186/s40814-022-01007-1. PMID 35227311